CLINICAL TRIAL: NCT03208439
Title: Interactive Cycling System Using Electromyography (EMG)-Driven Neuromuscular Electrical Stimulation (NMES) for Rehabilitation
Brief Title: Neuromuscular Electrical Stimulation Cycling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016.093-T
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG-driven NMES (Experimental): subjects will receive EMG-driven NMES cycling exercise.
  Interventions: Device: lower-limb cycling system
- passive pre-programmed NMES (Placebo Comparator): subjects will receive passive pre-programmed NMES during cycling exercise.
  Interventions: Device: lower-limb cycling system

INTERVENTIONS:
Device: lower-limb cycling system — patients will receive 30-minute cycling exercise

SUMMARY:
A new electromyography (EMG)-driven neuromuscular electrical stimulation (NMES)-cycling system is introduced to stroke survivors for lower-limb rehabilitation. The system will generate NMES to targeted muscle according to the user's voluntary intention, represented by the EMG signal during cycling.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of ischemic brain injury or intracerebral hemorrhage shown by magnetic resonance imaging or computed tomography after the onset of stroke;
2. sufficient cognition to follow simple instructions as well as understand the content and purpose of the study;
3. significant gait deficit (Functional Ambulatory Category, FAC, scale <4 [person cannot walk independently]).

Exclusion Criteria:

1. any additional medical or psychological condition that would affect their ability to comply with the study protocol, e.g., a significant orthopedic or chronic pain condition, major post-stroke depression;
2. severe hip, knee or ankle contracture that would preclude passive range of motion of the leg;
3. implanted cardiac device (e.g. pacemaker and internal defibrillator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Lower-Extremities Fugl-Meyer Assessment | 3-month follow up

SECONDARY OUTCOMES:
Elderly Mobility Scale | 3-month follow up
Berg Balance Scale | 3-month follow up
6-Minute Walking Test | 3-month follow up
10-Meter Walk Test | 3-month follow up
electroencephalography | 3-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kai-yu Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu C, Wang T, Leung KWC, Li L, Tong RK. Muscle Electrical Impedance Properties and Activation Alteration After Functional Electrical Stimulation-Assisted Cycling Training for Chronic Stroke Survivors: A Longitudinal Pilot Study. Front Neurol. 2021 Dec 15;12:746263. doi: 10.3389/fneur.2021.746263. eCollection 2021. PMID 34975713